CLINICAL TRIAL: NCT04547634
Title: Effect of a Telerehabilitation-exercise Intervention in Oncology Patients in the Covid-19 Pandemic
Brief Title: Telerehabilitation in Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher of CTS631 University of Malaga, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Teleclub_cam
Record Dates: First submitted 2020-08-17; First posted 2020-09-14 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-09

CONDITIONS: Cancer Metastatic; Cancer; Survivorship
Keywords: cancer; oncology; Metastasis; survivors; Exercise Therapy; Therapeutics; Complementary Therapies; covid-19
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; COVID-19 | interventions — Exercise Therapy; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The sample will receive of a Therapeutic Exercise and Education programme
  Interventions: Other: Therapeutic Exercise and Education
- Control (No Intervention): Subjects will be told to continue with their normal activity of daily living. After the intervention in the experimental group, the control group will be offered intervention.

INTERVENTIONS:
Other: Therapeutic Exercise and Education — The intervention will consist of 30 minutes of strength exercises followed by 20 minutes of endurance with aerobic training, individualized based on the evaluations of muscular strength and endurance. Sessions lasted 1 hour, carried out twice a week, for 12 weeks. This intervention will be complemented by nutritional education.
  Arms: Experimental

SUMMARY:
The aim is to analyze the feasibility and effect of an online Therapeutic Exercise and Education programme (TEEP) in cancer patient and survivors

DETAILED DESCRIPTION:
Current literature shows that Therapeutic Exercise has multiple benefits in oncology patients, such as improvements in function and quality of life, and ameliorates symptoms such as cancer-related fatigue. Furthermore, given the risk of obesity, both exercise and diet play a key role in recovery from cancer. In fact, current guidelines support the use of exercise with therapeutic purposes as a complement to cancer treatment.

As a consequence of the COVID-19 pandemic, oncology patients present more difficulties to attend programs, as the vast majority are immunosuppressed, and they are considered risk population. Therefore, new online (TEEP) must be developed to facilitate the benefits of these programs in the post-COVID Era. This study analyses the feasibility (in terms of suitability and verification of exercise prescription, absence and attendance type, and total days of attendance) and the effect (in weight, physical function, and symptoms) in cancer patients and survivors.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast patient, gynecological cancer patient, or breast cancer survivor under adjuvant treatment after surgical intervention.
* Having given informed consent to participate voluntarily in the program and to be in contact via telematics (email or messaging platform).
* Have a good internet connection
* Be accompanied by an adult on the day of assessment.
* Availability to access the computer on during the intervention.

Exclusion Criteria:

* Technophobia
* Domatophobia or self-report of adversity to be at home.
* Lack of logistical requirements (Internet and lack of skill in its use).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Suitability of exercise intensity | Through study completion, an average of 3 months
  Patients are asked before each session to mark in a numerical scale how are they feeling that day to push themselves and get their session well done. From 0 (very well) to 10 (very badly). Higher scores mean a worse feeling.
Verification of exercise intensity | Through study completion, an average of 3 months
  Patients are asked to score the feeling of perceived effort after the session with the Borg Perceived Exertion scale (6-20). Higher scores mean a worse perceived exertion.
Total attendance | After intervention, an average of 3 months
  Total of days of attendance
Absence type | Through study completion, an average of 3 months
  Reasons of absence, categorized as: personal matter, visit the oncology, medical appointment (no related to oncology treatment), health problem, connection problem or unknown.
Attendance type | Through study completion, an average of 3 months
  Attendance type, categorized as: full attendance, partly attendance because of lack of time, partly attendance because of internet connection problem

SECONDARY OUTCOMES:
Change from Cancer-Related Fatigue (CRF) | Prior and after intervention, an average of 3 months
  The Spanish version of the Piper Fatigue Scale-Revised (PFS-R) will be used. Its total score is the sum of all items (from 0 to 220), with higher values indicate a higher level of fatigue (worse outcome)
Change from Functional capacity | prior and after intervention, an average of 3 months
  It will be tested by 30-second Sit-To-Stand Test (30-STS), number of repetitions completed.
Change from Upper limb functionality (%) | prior and after intervention, an average of 3 months
  the Spanish version of Upper Limb Functional Index (ULFI) questionnaire will be filled online
Change from Lower limb functionality (%) | prior and after intervention, an average of 3 months
  the Spanish version of Lower Limb Functional Index (LLFI) questionnaire will be filled online
Change from Quality of life (self-reported questionnaire) | prior and after intervention, an average of 3 months
  It will be assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0. EORTC QLQ-C30 comprises 30 items and contains five functional scales, three symptom scales, a global health status/QoL scale, and six single items. Raw scores can be linearly converted to a 0-100 scale with higher scores reflecting higher levels of function (better outcome) and higher levels of symptom show bigger problems (worse outcome).
Change from specific Breast Cancer Quality of life (self-reported questionnaire) | prior and after intervention, an average of 3 months
  It will be assessed by The European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life questionnaire (EORTC QLQ-BR23). This is a breast cancer module of EORTC QLQ-C30 which contains 23 items that assess disease symptom, side effects of treatment, body image, sexual functioning, and future perspective. All items are rated on a 4-point scale (from 1- not at all, to very much). Higher scores represent better functioning (better outcome), and higher scores of symptom show bigger issues (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cuesta Vargas, Málaga, Spain